CLINICAL TRIAL: NCT00323141
Title: Prospective Randomized Trial to Study the Effectiveness of an Intraperitoneal Mesh With an Overlap of 3cm Versus a Rives-Stoppa Repair With an Overlap of 6cm With Patients With a Hernia Umbilicalis
Brief Title: Intraperitoneal Mesh With 3cm Overlap Versus a Rives-Stoppa Repair With a 6cm Overlap in Hernia Umbilicalis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/079
Record Dates: First submitted 2006-05-07; First posted 2006-05-09 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Hernia, Umbilical
Keywords: Hernia umbilicalis
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ventralex (Active Comparator)
  Interventions: Device: Ventralex versus Leight Weight Vypro II prothesis
- Leight Weight Vypro II prothesis (Active Comparator)
  Interventions: Device: Ventralex versus Leight Weight Vypro II prothesis

INTERVENTIONS:
Device: Ventralex versus Leight Weight Vypro II prothesis — Ventralex and Leight Weight Vypro II prothesis are compared.

SUMMARY:
To study the advantages and disadvantages of a Ventralex prothesis versus Light Weight Vypro II prothesis in patients with a hernia umbilicalis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic hernia umbilicalis
* > 18 years old

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03-11 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Number of relapses after 1 and 3 years | after 1 and 3 years

SECONDARY OUTCOMES:
Duration of surgery | Depends from type of surgery.
Duration of hospitalisation | Depends from type of surgery.
Frequency of complications | After 1 and 3 years.
Pain assessment | After 1 and 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be